CLINICAL TRIAL: NCT06171334
Title: Open-label, Single-center, Single-arm Futility Trial Evaluating Daily Remote Ischemic Conditioning for Reducing Progression of Disability in Patients With Primary Progressive Multiple Sclerosis (PPMS)
Brief Title: Remote Ischemic Conditioning in PPMS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REB23-1062
Record Dates: First submitted 2023-11-27; First posted 2023-12-14 (Actual); Last update posted 2024-05-09 (Actual); Status verified 2023-11

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: This is a phase II open-label, single-center, single-arm futility trial. The study will follow the Simon-2-stage MiniMax design for futility studies.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- RIC (Experimental)
  Interventions: Device: Remote ischemic conditioning

INTERVENTIONS:
Device: Remote ischemic conditioning — The intervention consists in Remote Ischemic conditioning (RIC), one session of 40-minutes duration per day for 12 months. The procedure will be performed by using an electric auto-control device by SnapDx Inc (Calgary, Canada) with a blood pressure cuff that inflates up to a pressure of 200 mmHg during the ischemic period. Participant will self-administer the RIC procedure at their home. The device records and documents each RIC cycle.

SUMMARY:
Progressive MS remains the most difficult therapeutic challenge. Remyelination is a promising therapeutic strategy but an effective pharmacologic intervention remains elusive. Remote ischemic conditioning (RIC) is a non-pharmacologic intervention that has been studied in the context of stroke, where transient limb ischemia leads to neuroprotection. However, RIC has not yet been studied in MS. The investigators hypothesized that repeating RIC over several days may induce molecular/cellular changes in the CNS that promote remyelination. Since RIC is safe, tolerable and ready for clinical translation (recent stroke trials have shown promise), the investigators will run a clinical study to test RIC in people with primary progressive MS.

The purpose of this clinical trial is to determine if RIC in a dose of 4 cycles daily can prevent worsening of walking ability in people PPMS. The trial is funded through MS Canada as well as a private donation to the Hotchkiss Brain Institute MS Translational Clinical Trials Research Program and the University of Calgary. There is no sponsorship from the pharmaceutical industry.

DETAILED DESCRIPTION:
Remote Ischemic conditioning (RIC): Ischemic-preconditioning entails inducing short periods of cyclical tissue ischemia that confers subsequent protection against ischemia-reperfusion-injury. The rationale is that short periods of ischemia do not cause irreversible injury, but instead induce an endogenous protective environment. This short period of ischemia is not injurious, and it triggers endogenous protective signals (such as anti-inflammatory and antioxidant molecules) that reach distant organs, such as the heart, liver or the CNS. As an endogenous, non-specific response, the mechanisms involved in RIC are complex and include inflammation, oxidative stress, changes in endothelial function, cell survival etc.

Current treatments for progressive Multiple Sclerosis (the immune-modulators Siponimod and Ocrelizumab) are only modestly effective and primarily benefit people with active inflammatory disease activity (recent relapses and/or enhancing lesions on MRI). Progression free of inflammatory activity is characterized by slow accumulation of disability, greatly affecting quality of life in people with Multiple Sclerosis (MS). The investigators believe RIC is ideally suited to be tested as a therapy for progression in MS. Recent clinical trials in vascular disease have shown that daily RIC can be performed for up to a year and suggested an all-cause mortality benefit. In a recent (RICAMIS trial, 2022) multicenter, randomized trial of people with acute ischemic stroke (> 1,000 participants), 14-day RIC treatment led to improved functional outcomes at 6-months. No serious side effects were reported, and tolerability was good.

This important study was the first phase III trial to find a "protective" effect for RIC in neurological disease, and highlights the timeliness and potential for re-purposing RIC as a therapy for MS.

In this trial, the investigators will investigate whether RIC treatment can prevent disability worsening in people with Primary Progressive MS (PPMS).

The primary objective of this trial is to demonstrate non-futility of RIC for reducing progression of disability, as measured with the timed 25-foot walk (T25FW), in people with PPMS.

This is a phase II open-label, single-center, single-arm futility trial. The study will follow the Simon-2-stage MiniMax design for futility studies.

ELIGIBILITY:
Inclusion Criteria:

Written informed consent obtained

* Men and women aged of 18 and 65 years inclusive
* With Primary Progressive Multiple Sclerosis, according to current diagnostic criteria
* Screening Expanded Disability Status Scale score between 4.0 and 6.5 inclusive
* Screening timed 25-foot walk (average of two trials) of 5.5 seconds or more

Exclusion Criteria:

Patients whose screening MRI scan shows gadolinium enhancing lesions

* Patients with known renal insufficiency
* Patients with known significant hepatic impairment
* Patients with known allergy to gadolinium MRI contrast agent
* Patients currently using immune-modulators such as ocrelizumab or hydroxychloroquine
* Patients currently using therapeutic anticoagulation (blood thinners, such as warfarin, apixaban, rivaroxaban, dabigatran, enoxaparin)
* Patients currently using Fampridine or 4-aminopyridine
* Patients planning to start Fampridine or 4-aminopyridine during the study period
* Patients planning to start Baclofen or Tizanidine during the duration of the study
* Patients who increase the dose of Baclofen or Tizanidine during the study period
* Patients who receive treatment with Botulinum toxin in the leg muscles during the study period
* Patients who are unable or unwilling to undergo gadolinium enhanced MRI scans
* Patients with known history of thrombotic events in the upper extremities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2024-07-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Timed 25-foot walk | 12 MONTHS
  The primary endpoint in this study will be the worsening of disability, defined as an increase by 20% or more in the timed 25-foot walk (average of two trials) at 12 months follow-up compared to baseline.

SECONDARY OUTCOMES:
Nine Hole Peg Test | 12 MONTHS
  A validated test of upper limb motor function. Increased times (longer time to finish test). indicates worse function. A 20% change is considered significant.
MRI measure of remyelination | 12 MONTHS
  MRI will be done at baseline and at 12-months. Normal appearing white matter Diffusion Tensor Imaging. Provides a numeric value, whew higher values indicate "improved" myelin integrity. The investigators will test changes in this MRI measure over time.
SDMT (Single digit modalities test) | 12 MONTHS
  A validated test of processing speed (an aspect of cognition). Lower numbers indicate worse processing speed. An 8-point change is considered significant.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Canada

IPD SHARING:
Plan to Share IPD: Yes
De-identified data may be shared to qualified researchers, upon reasonable request, after the end of study and primary data analysis.
Supporting Information: Study Protocol, Analytic Code
Time Frame: After end of study and data analysis

REFERENCES:
- [Background] Chen HS, Cui Y, Li XQ, Wang XH, Ma YT, Zhao Y, Han J, Deng CQ, Hong M, Bao Y, Zhao LH, Yan TG, Zou RL, Wang H, Li Z, Wan LS, Zhang L, Wang LQ, Guo LY, Li MN, Wang DQ, Zhang Q, Chang DW, Zhang HL, Sun J, Meng C, Zhang ZH, Shen LY, Ma L, Wang GC, Li RH, Zhang L, Bi C, Wang LY, Wang DL; RICAMIS Investigators. Effect of Remote Ischemic Conditioning vs Usual Care on Neurologic Function in Patients With Acute Moderate Ischemic Stroke: The RICAMIS Randomized Clinical Trial. JAMA. 2022 Aug 16;328(7):627-636. doi: 10.1001/jama.2022.13123. PMID 35972485
- [Background] Camara-Lemarroy CR, Metz L, Smith EE, Dunn JF, Yong VW. Expanding the Potential Therapeutic Options for Remote Ischemic Preconditioning: Use in Multiple Sclerosis. Front Neurol. 2018 Jun 19;9:475. doi: 10.3389/fneur.2018.00475. eCollection 2018. No abstract available. PMID 29971043